CLINICAL TRIAL: NCT02139501
Title: A Randomized Study to Evaluate the Efficacy and Safety of Different Doses and Frequencies of Recombinant Human Thrombopoietin (rhTPO) in the Management of Primary Immune Thrombocytopenia (ITP)
Brief Title: An Investigation of rhTPO With Different Frequencies in the Management of ITP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: The First Affiliated Hospital of Dalian Medical University (Other); Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITP-Thrombopoietin
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2014-11

CONDITIONS: Immune Thrombocytopenia
Keywords: Recombinant Human Thrombopoietin; Dose and frequency; Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Thrombopoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- rhTPO, 300Units/kg ,daily for 14 consecutive days (Experimental): 10 enrolled patients randomly receive rhTPO at a dose of 300Units/kg ,daily for 14 consecutive days
  Interventions: Drug: Recombinant Human Thrombopoietin (rhTPO)
- rhTPO, 300Units/kg ,one times every other day for 7 times (Experimental): 10 enrolled patients randomly receive rhTPO at a dose of 300Units/kg ,one times every other day for 7 times.
  Interventions: Drug: Recombinant Human Thrombopoietin (rhTPO)
- rhTPO, 300Units/kg ,daily for 7 consecutive days (Experimental): 10 enrolled patients randomly receive rhTPO at a dose of 300Units/kg ,daily for 7consecutive days.
  Interventions: Drug: Recombinant Human Thrombopoietin (rhTPO)

INTERVENTIONS:
Drug: Recombinant Human Thrombopoietin (rhTPO) — rhTPO was given intravenously at a dose of300Units/kg ,daily for 14 consecutive days;at a dose of 300Units/kg ,one times every other day for 7 times; or at a dose of 300Units/kg ,daily for 7 consecutive days
  Other Names: tpiao; Recombinant Human Thrombopoietin; Recombinant Human TPO

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University and other well-known hospitals in China. In order to study the efficacy and safety of different dose and frequency Recombinant Human thrombopoietin in treating the primary immune thrombocytopenia (ITP)

DETAILED DESCRIPTION:
The investigators are undertaking a parallel group, multicentre, randomised controlled trial of 30 primary ITP adult patients from 3 medical centers in China. They will be randomly assigned in a 1:1:1 ratio into three groups .The patients in group A (total 10 patients) will receive rhTPO at a dose of 300Units/kg ,daily for 14 consecutive days;The patients in group B will receive rhTPO at a dose of 300Units/kg ,one times every other day for 7 times.The patients in group C will receive rhTPO at a dose of 300Units/kg ,daily for 7 consecutive days .All the patients will follow with a flexible dosage depending on platelet count during the following 12 weeks.

Platelet counts, bleeding and other symptoms were evaluated before and after treatment, in order to evaluate the efficacy and safety of different dose and frequency Recombinant Human thrombopoietin in treating the primary immune thrombocytopenia (ITP)

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years old, may be male or female.
2. Diagnosed with ITP meeting the diagnostic criteria for immune thrombocytopenia.
3. Patients who have no response or relapsed after Corticosteroid.
4. To show a platelet count < 30×10^9/L, and with bleeding manifestations.
5. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit.
2. Received second-line ITP-specific treatments (eg, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) within 3 months before the screening visit.
3. Received high-dose steroids or IVIG in the 3 weeks prior to the start of the study.
4. Current HIV infection or hepatitis B virus or hepatitis C virus infections.
5. Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)
6. Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period.
7. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.
8. Patients who are deemed unsuitable for the study by the investigator .

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Early Response | 14 days
  response rate (CR+R) at the 14th day and the 14th week from the initial injection of rhTPO. CR is defined as platelet count ≥ 100×10^9/L, and R is defined as platelet count of >30 × 10^9/L with a least a doubling of the baseline value.

SECONDARY OUTCOMES:
Safety | 1 years
  The type and frequency of therapy associated adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, Dr, Principal Investigator — Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China